CLINICAL TRIAL: NCT07402408
Title: Comparison of Band Tissue Flossing Method and Traditional Cuff Method for Blood Flow Restriction Training in Patients With Knee Osteoarthritis
Brief Title: Blood Flow Restriction Training in Knee Osteoarthritic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS/REC/MS-PT/02171
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthristis
Keywords: Blood flow restriction therapy; Knee Osteoarthritis; Range of Motion
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction with Floss band (group A) (Experimental): seated knee extension and knee press while floss band is tied at proximal thigh.
  Interventions: Other: Blood flow restriction training with Floss band
- Blood flow restriction with pneumatic cuff (group B) (Experimental): seated knee extension and knee press exercises with pneumatic cuff tied at proximal thigh
  Interventions: Other: Blood flow restriction training with pneumatic cuff

INTERVENTIONS:
Other: Blood flow restriction training with Floss band — seated knee extension exercise and knee press exercises (4 sets; repetitions: 30,15,15,15) performed for four weeks with three sessions per week. Exercises performed with 20% of one repetition maximum. Floss band was tied at proximal thigh with 50% stretch in proximal to distal direction starting from above the patella and moving towards groin.
  Arms: Blood flow restriction with Floss band (group A)
Other: Blood flow restriction training with pneumatic cuff — seated knee extension exercises and knee press exercises (4 sets; repetitions: 30,15,15,15) performed for four weeks with three sessions per week. Exercises performed with 20% of one repetition maximum. Clinical cuff was tied at proximal thigh with 40% of limb occlusion pressure.
  Arms: Blood flow restriction with pneumatic cuff (group B)

SUMMARY:
The aim of this study was to compare the effect of band tissue flossing method and traditional cuff method for blood flow restriction training on pain, range of motion, muscle strength and functional status in patients with knee osteoarthritis. Symptoms of this condition limit patient's ability to perform high load strengthening. Blood flow restraining training allows strengthening with lower loads. 46 subjects were divided in two groups, 23 subjects in each group. knee extension and knee press exercises were performed. In group A floss band was tied on thigh and in group B pneumatic cuff was applied on thigh. 40-60 years individual with knee osteoarthritis were included. outcome measures were assessed at baseline, after 1st session, after 2nd week and after 4th week.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disorder affecting 528 million people worldwide. It occurs in individuals of age 40 years and above. Most affected joint is knee with prevalence of 60%-85% of total OA cases being 1.39 times higher in women than men. It is characterized by progressive damage to articular cartilage, leading to pain, stiffness, and reduced mobility negatively impacting function and quality of life of affected patients.

Obesity, low level of physical activity, joint overload, muscle imbalance in the knee joint, reduced weight and muscle strength in the lower limbs are the factors which can be modified. Quadriceps strengthening is considered as a first-line therapy making resistance training a common practice in OA management.

A useful alternative to high intensity exercises which are not tolerable by osteoarthritic patients is blood flow restriction (BFR) training. In BFR a cuff is applied around the proximal aspect of the affected limb, causing partial arterial and full venous occlusion, thereby inducing localized hypoxia and the accumulation of metabolites, imitating the effects of high load resistance training without using heavy load and higher repetition. BFR reduces pain along with improving muscle strength, and function in patients with osteoarthritis (OA) and rheumatoid arthritis.

The tissue flossing technique is also called BFR or Kaatsu training. The use of tissue flossing (TF) is a relatively recent treatment modality that gained popularity through the book by Starrett and Cordoza. The mechanisms involved in TF are similar to ischemic preconditioning or BFR training in which an application of an external pressure is used, above or below the muscle or joint, with the application of a tourniquet/inflatable cuff in the most proximal portion of the limb in the case of BFR or an elastic band. Tissue flossing can improve the range of motion or performance, speed up recovery, and decrease the pain caused by various diseases or injuries. The intervention consists of wrapping tissue flossing band around a body region (joint or soft-tissue) using a 50% overlapping in circumferential pattern (distal to proximal), with a relative stretch ranging from 50-75% of the band maximal length, and a treatment duration ranging from 2 minutes to 6 minutes or exercise repetition range from 10 to 30 repetitions.

In 2015, research evaluated effects of BFR on older women and concluded that addition of BFR with resistance training significantly increased leg press or quadriceps strength in older women.

In 2018, a study included forty-eight women with knee OA who were randomized into three groups: low intensity training with BFRT, low intensity training with partial BFRT, and high-intensity resistance training. BFRT and HI-RT were similarly effective in increasing muscle strength, quadriceps muscle mass, and functionality in knee OA patients. Importantly, BFRT was also able to improve pain while inducing less joint stress, emerging as a feasible and effective therapeutic adjuvant in OA management In 2023, study concluded that Low-intensity resistance training with and without blood flow restriction was similarly effective in enhancing functional status in subjects with knee osteoarthritis. A pilot study performed in 2024 on older adults with knee OA shows that (BFR) significantly reduced pain. In the timed up and go and sit to stand tests, completion times were significantly reduced. Thigh and calf circumferences, as well as thigh muscle thickness significantly increased after exercise. However, isokinetic knee strength did not show significant changes. RCT performed in 2024 investigated the long-term effects of BFRT in patients with knee OA and concluded that BFRT is a promising tool to optimize patient outcomes in the rehabilitation of KOA in the long term.

A study in 2021 concluded that compared to the control condition, the flossing treatment showed a positive effect on the maximum voluntary contraction of the knee extensors .

Another study in 2020 states, flossing yielded greater improvements in the passive knee extension test and yielded significant improvements in the maximal eccentric knee extension contraction than dynamic stretching flossing on hamstring muscles is more beneficial than dynamic stretching with respect to increasing ROM and muscle exertion.

A study in 2021 concluded that floss band intervention can significantly improve the flexibility of the quadriceps and hamstrings, quadriceps muscle force output, and dynamic balance without impeding knee proprioception.

According to another study in 2020, flossing bands caused a reduction in perceived knee pain and improved vertical jump performance in young male recreational athlete.

A study in 2022 compared flossing and pneumatic cuff for evaluating their hemodynamic responses to blood flow restriction in healthy population. They concluded that floss band can cause blood flow restriction similar to pneumatic cuff. Clinical application of floss band in KOA population remains underexplored.

To date, no randomized controlled trial has directly compared therapeutic effects of these two BFR interventions in knee OA patients creating a gap in literature. Therefore, the significance of this study lies in its potential to explore the clinical effectiveness of both methods. By doing so, the findings might help inform future research or clinical protocols regarding the use of practical BFR methods in knee OA rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Pain more than or equal to 3 on NPRS
* Range of motion ≤ 100-degree flexion and ≤ 0-degree extension
* Those who have knee osteoarthritis, according to KL (Grade 1 and 2)
* Genders: Male and Female

Exclusion Criteria:

* Cardiovascular condition e.g., hypertension, thromboembolism, lymphatic diseases etc.
* Muscle/tendon/ ligament injuries
* Any surgery, skin infection, trauma, pregnancy, fracture and fall
* Patient with intra articular steroidal therapy with in last 6 months
* Patient unwilling to participate and comply with the study session

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-24 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  Changes from baseline were assessed using NPRS scale. It is a one-dimensional measure of pain severity in adults including those suffering from chronic pain. Scale has ratings of 0 to 10, with higher points indicating higher levels of pain severity. it is a valid tool for assessing pain in knee OA patients.

SECONDARY OUTCOMES:
Knee Flexion Range of motion | 4th week
  Changes in knee flexion range of motion from baseline were assessed using universal goniometer. Goniometer is the most common instrument utilized for measuring available range of motion. Universal Goniometer Comes in two variations one is short arm whereas one is long arm. The one with short arm is used for smaller joints like the wrist, elbow, or ankle. On the other hand, long arm goniometers provide greater accuracy for knee and hip joints which have long bones acting as levers
Knee Extension Range of Motion | 4th week
  Changes from baseline in knee extension range of motion were assessed with goniometer. It is the most common instrument utilized for measuring available range of motion. Universal Goniometer Comes in two variations one is short arm whereas one is long arm. The one with short arm is used for smaller joints like the wrist, elbow, or ankle. On the other hand, long arm goniometers provide greater accuracy for knee and hip joints which have long bones acting as levers
Quadriceps strength (dynamometer) | 4th week
  Quadriceps muscle strength changes from baseline were assessed using crane scale dynamometer. Participant sits in chair with hips and knees flexed to 90 degrees. The hook of dynamometer is secured to the ankle with a strap, while from behind the dynamometer is fixed to leg of chair to provide a stable anchor. As the participant performs knee extension the force generated is recorded in newtons or kilograms. It is a valid and reliable tool for assessing strength of knee extensors.
Western Ontario and McMaster Universities (WOMAC) index | 4th week
  WOMAC index was developed in order to fill the need for an outcome instrument that could be responsive to change in OA-related symptoms following a clinical trial. It includes five questions about pain, two about stiffness, and seventeen on degree of disability of activities of daily living. total score is converted to percentage. higher scores mean severe symptoms.
30 Second Sit to Stand Test (STS) | 4th week
  The 30 Second Sit to Stand Test (STS) is also known as 30 Second Chair Stand Test (30CST), was initially designed for testing leg strength and endurance in older adults. It is used for adults of 18-64 years, older adults (65 years and above), and people with osteoarthritis. A person stands up and sits down five times as quickly and safely as possible, with their arms folded across their chest, A longer time indicates weaker leg strength and a greater risk of falls. It records the number of times a person can sit and stand within 30 seconds
Timed Up and Go Test (TUG) | 4th week
  This test is for assessing ambulatory transition in knee OA patients. For this test participant stands from armed chair, walks with comfortable pace to a line 3 m away, at end point turns, and returns to sitting position in chair. Participant can't use walking aid during task. Time is recorded in which task is done.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Institute of Medical Sciences (P.I.M.S.), Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No